CLINICAL TRIAL: NCT06007066
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled Phase II Study of The Efficacy And Safety of HSK16149 In The Treatment of Patients With Orthopedic Perioperative Analgesia
Brief Title: HSK16149 for Perioperative Analgesia in Orthopedic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK16149-204
Record Dates: First submitted 2023-03-05; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Preoperative administration of HSK16149 40mg (Experimental): HSK16149 40mg will be administered the night before and 2h before surgery
  Interventions: Drug: HSK16149 capsule
- Preoperative administration of HSK16149 60mg (Experimental): HSK16149 60mg will be administered the night before and 2h before surgery
  Interventions: Drug: HSK16149 capsule
- Preoperative and postoperative administration of HSK16149 40mg (Experimental): HSK16149 40mg will be administered orally the night before surgery, 2h before surgery, 4h and 16h after surgery
  Interventions: Drug: HSK16149 capsule
- Preoperative and postoperative administration of HSK16149 60mg (Experimental): HSK16149 60mg will be administered orally the night before surgery, 2h before surgery, 4h and 16h after surgery
  Interventions: Drug: HSK16149 capsule
- placebo (Placebo Comparator): The placebo will be administered orally the night before surgery, 2h before surgery, 4h and 16h after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK16149 capsule — Subjects will be given 40mg or 60mg of HSK16149 orally.
  Other Names: HSK16149
  Arms: Preoperative administration of HSK16149 40mg; Preoperative administration of HSK16149 60mg; Preoperative and postoperative administration of HSK16149 40mg; Preoperative and postoperative administration of HSK16149 60mg
Drug: Placebo — Subjects will be given HSK16149 placebo orally.
  Other Names: HSK16149 placebo
  Arms: placebo

SUMMARY:
This study will compare the effect and safety of HSK16149 with placebo on perioperative analgesia in orthopedic surgery, and explore the dosage of HSK16149 capsules for orthopedic analgesia during perioperative period.

DETAILED DESCRIPTION:
This study included patients who have orthopedic surgery under general anesthetic, with expected operation time ≤4h.

Subjects were given 40mg or 60mg of HSK16149 or placebo orally the night before surgery, 2h before surgery, 4h and 16h after surgery, for a total of 4 times during the whole treatment period.

Subjects will receive intravenous patient-controlled analgesia (PCA) morphine for pain in the immediate postoperative period. If PCA is insufficient, rescue analgesia of morphine may be given I.V. as determined by the investigator.

After the treatment period, the subjects will be followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 75 years (included);
2. Elective orthopedic surgery under general anesthesia, expected operation time ≤4 hours and postoperative morphine analgesia time ≥24 hours;
3. 18kg/m^2≤BMI≤30 kg/m^2;
4. American Society of Anesthesiologists (ASA) grade I and II;

Exclusion Criteria:

1. Any of the following medical histories or conditions prior to screening:

   * Long history of chronic pain;
   * history of severe cardiovascular or respiratory disease;
   * history of neurological or psychiatric disorders;
   * history of acute poisoning with alcohol, hypnotics, analgesics or other drugs acting on the central nervous system;
   * major surgery within 3 months;
   * patients with high bleeding risk;
   * history of renal disease treated with dialysis within 28 days before surgery;
   * have active infection within the past 2 weeks;
2. Use of any of the following medications or treatments:

   * opioid analgesics for more than 10 consecutive days within 3 months prior to screening;
   * other analgesics before randomization if the last dose was taken less than 5 half-lives of the drug (according to the label);
3. Abnormal laboratory tests during screening:
4. Hypertension that is not adequately controlled by antihypertensive drugs (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg), or systolic blood pressure ≤90 mmHg during screening;
5. A history of drug abuse, and/or alcohol abuse in the 3 months prior to screening;
6. Participated in another clinical trial and received IMP within 30 days prior to screening;
7. Pregnant or lactating women;
8. Unwillingness to use reliable contraceptive methods from the time of screening until 28 days after the last dose of IMP;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Morphine Consumption | Participants received PCA pump, an average of 24 hours after surgery
  IV Patient Controlled Analgesia (PCA) morphine for pain management in the immediate postoperative period for an average of 24 hours after surgery. If PCA is insufficient, rescue analgesia of morphine may be given I.V. as determined by the investigator.
  Total morphine consumption = PCA morphine consumption + rescue analgesia morphine consumption.

SECONDARY OUTCOMES:
NRS at rest and during exercise | 1, 2, 6, 12, 18, and 24 hours after surgery
  NRS:0 (no pain) to 10 (worst possible pain)
Time of first rescue analgesia with morphine after surgery | Within 24 hours after surgery
Incidence of adverse reactions associated with morphine | Within 24 hours after surgery
The frequency of rescue analgesia with morphine | Within 24 hours after surgery
The total number of PCA presses and the number of effective PCA presses | Within 24 hours after surgery
Daily Sleep Interference Scale (DSIS) | Within 24 hours after surgery
  Subjects review their sleep status during the past 12 hours at 8:00 a.m. on the day of surgery.
  DSIS: 0 (not affecting sleep) to 10 (unable to sleep)
Subjects analgesic satisfaction score | Within 24 hours after surgery
  Analgesic satisfaction score: 0 (not satisfied) to 10 (very satisfied)
Investigators analgesic satisfaction score | Within 24 hours after surgery
  Analgesic satisfaction score: 0 (not satisfied) to 10 (very satisfied)
Number of participants with treatment-related adverse events(TEAE) as assessed by CTCAE v5.0. | From enrollment to 72 hours after surgery
  Number and severity of AEs, clinical laboratory abnormalities, physical examinations, 12-lead electrocardiograms (ECGs)(including QT Interval,QTc Interval and PR Interval), and vital signs.

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Foshan Fuxing Chancheng Hospital, Foshan, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Beijing Jishuitan Hospital Guizhou Hospital, Guiyang, Guizhou
  - Zunyi University Affiliated Hospital, Zunyi, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Xiangya Third Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of South China University, Hengyang, Hunan
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Chengdu Third People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Guangyuan First People's Hospital, Guangyuan, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Sino-Japanese Friendship Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No